CLINICAL TRIAL: NCT04467515
Title: A Multi-Center Open Label Dose Escalation and Dose Expansion Study to Evaluate Safety, Tolerability, Dosimetry, and Preliminary Efficacy of the HER2 Directed Radioligand CAM-H2 in Patients With Advanced/Metastatic HER2-Positive Breast, Gastric, and GEJ Cancer
Brief Title: A Study to Evaluate Safety, Tolerability, Dosimetry, and Preliminary Efficacy of the HER2 Directed Radioligand CAM-H2 in Patients With Advanced/Metastatic HER2-Positive Breast, Gastric, and Gastro-Esophageal Junction (GEJ) Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per Strategic Sponsor decision
Sponsor: Precirix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAMH2_1001
Record Dates: First submitted 2020-06-10; First posted 2020-07-13 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Advanced/Metastatic HER2-positive Breast, Gastric, Gastroesophageal Junction Cancer With Disease Progression Following Anti-HER2 Standard of Care Treatment

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2 multi-center, open label, dose escalation and dose expansion study to evaluate safety, tolerability, dosimetry, PD, and efficacy of the targeted radionuclide therapeutic CAM H2 in patients with progressive, advanced/metastatic HER2 positive breast, gastric, and GEJ cancer with disease progression following anti-HER2 standard of care treatment. The study is comprised of a Treatment Period, consisting of a maximum of 4 cycles (12 weeks per cycle) of study drug, and a Long Term Follow Up Period.
  The study will be comprised of the following:
  * Dose Escalation Phase Followed by a Long Term Follow Up (LTFU) period
  * Dose Expansion Phase Followed by a LTFU period
  In the dose expansion phase of the study, the patients will be given the recommended dose for Phase 2 (RDP2) determined in the dose escalation phase. Similar to the dose escalation phase, all patients will receive at least 1 cycle of CAM-H2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): The dose escalation phase of the study will be an open label 3 + 3 design, where at least 3 patients are treated at each dose level. Dose escalation will be done via increases of the nominal activity of CAM-H2 in cohorts of 3 to 6 patients.
  In the dose expansion phase of the study, the patients will be given the RDP2 determined in the dose escalation phase. Similar to the dose escalation phase, all patients will receive at least 1 cycle of CAM-H2.
  Interventions: Drug: CAM-H2

INTERVENTIONS:
Drug: CAM-H2 — All patients will receive at least 1 cycle of CAM-H2. Patients with CB may receive 4 cycles of CAM-H2, each cycle given as 2 IV administrations, 4 weeks apart.

SUMMARY:
This is a Phase 1/2 multi-center, open label, dose escalation and dose expansion study to evaluate safety, tolerability, dosimetry, pharmacodynamics (PD), and efficacy of the targeted radionuclide therapeutic CAM-H2 in patients with progressive, advanced/metastatic HER2-positive breast, gastric, and GEJ cancer with disease progression following anti-HER2 standard of care treatment.

DETAILED DESCRIPTION:
The study duration for each phase will be up to 18 months. The study is comprised of a Treatment Period, consisting of a maximum of 4 cycles (12 weeks per cycle) of study drug, and a 12-month Long-Term Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed voluntarily before any study-related procedure is performed, indicating that the patient understands the purpose of, and procedures required for, the study and is willing to participate in the study;
2. Males and females ≥ 18 years of age at screening;
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1;
4. HER2-positive locally advanced or metastatic breast cancer refractory to standard cancer treatment or HER2-positive locally advanced or metastatic gastric or GEJ cancer, refractory to standard cancer treatment.
5. Patients should have a minimum of 1 measurable lesion as defined by RECIST version 1.1 or a minimum of 1 measurable lesion as defined by RANO-BM within 4 weeks of the first dose of the study drug (Day 1). The lesion has to be a new lesion or progression of an existing lesion under the current therapy.
6. Any previous anti-HER2 treatment for advanced or metastatic disease is allowed. Patients with breast cancer should have had at least 2 previous systemic anticancer treatments for recurrent, locally advanced or metastatic cancer. Patients with gastric cancer or GEJ cancer should have had at least 1 previous anti-HER2 treatment.
7. Life expectancy > 6 months;
8. Adequate organ function, determined by the following laboratory tests:

   * Adequate kidney function with an estimated glomerular filtration rate (eGFR) of >59 mL/minute calculated using the Chronic Kidney Disease Epidemiology Collaboration equation;
   * Adequate hepatic function defined as an alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x the upper limit of normal (ULN), or <5 x ULN in patients with liver metastases, and total bilirubin <2 x ULN;
   * Neutrophil count >1500 cells/mm3 without growth factor support (14 days after last PEGylated granulocyte colony stimulating factor or 7 days after regular granulocyte colony stimulating factor);
   * Platelet count >100,000 cells/mm3 without platelet transfusion in the last 2 weeks;
   * Hemoglobin >9.0 g/dL without blood transfusion in the last 2 weeks; and
   * Adequate coagulation defined as an international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time <1.5 x the upper limit of the institutional normal range;
9. Baseline left ventricular ejection fraction ≥ 50% as measured by echocardiography or multigated acquisition scan.
10. Absence of any psychological, family, sociological, or geographical circumstance that could potentially represent an obstacle to compliance with the study protocol and the follow-up schedule, as determined by the Investigator. These circumstances will be discussed with the patient before enrollment in the study; and
11. Female patients of childbearing potential (ie, ovulating, premenopausal, and not surgically sterile) must have a negative pregnancy test at screening and prior to study drug administration. Patients and their partners of childbearing potential must be willing to use 2 methods of contraception, 1 of which must be a barrier method, for the duration of the study and until 6 months after study drug administration. Medically acceptable barrier methods include condom with spermicide or diaphragm with spermicide. Medically acceptable non-barrier contraceptive methods include intrauterine devices or hormonal contraceptives (oral, implant, injection, ring, or patch).

Exclusion Criteria:

1. Presence of frank leptomeningeal disease as a unique central nervous system feature or in association with brain parenchymal measurable lesion(s);
2. Symptomatic brain metastases; Note: Patients with asymptomatic treated and untreated brain metastases are eligible.
3. Previous local therapy for brain metastases, such as neurosurgery, stereotactic radiotherapy, or whole brain radiotherapy, administered within 6 weeks prior to administration of CAM-H2; Note: Previous therapy for brain metastases administered at least 6 weeks prior to CAM-H2 administration will be allowed.
4. For patients with brain metastases, any increase in corticosteroid dose during the 4 weeks prior to the first administration of CAM-H2.

   Note: Corticosteroid treatment in a stable dose or decreasing dose for at least 4 weeks prior to the first administration of CAM-H2 is allowed.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics or psychiatric illness/social situations that would limit compliance with study requirements;
6. Uncontrolled thyroid disease, defined as free triiodothyronine (T3) and free thyroxine (T4) > 3 x ULN at screening;
7. Uncontrolled diabetes defined as a fasting serum glucose > 2 x ULN or glycated hemoglobin levels > 8.5% at screening;
8. Gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (eg, Crohn's, ulcerative colitis);
9. Current active hepatic or biliary disease (exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per Investigator assessment);
10. Ongoing peripheral neuropathy of Grade > 2 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0;
11. Severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

    * Symptomatic congestive heart failure of New York Heart Association Class III or IV;
    * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease; or
    * Liver disease, including cirrhosis and severe hepatic impairment;
12. Active (acute or chronic) or uncontrolled severe infections;
13. Known history of HIV, hepatitis B, or active hepatitis C virus at screening;
14. Prior investigational anticancer therapy within 4 weeks prior to the first administration of CAM-H2.
15. Patients who have had a major surgery or significant traumatic injury within 4 weeks prior to the first administration of CAM-H2, who have not recovered from side effects of any major surgery (defined as requiring general anesthesia), or have a major surgery planned during the course of the study;
16. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin or stage I uterine cancer;
17. Radiation therapy for metastatic disease foci outside the brain, administered within 3 weeks prior to the first administration of CAM-H2;
18. Known hypersensitivity to any of the study drugs (including inactive ingredients), including iodine allergy;
19. History of significant comorbidities that, in the Investigator's judgement, may interfere with study conduct, response assessment, or informed consent;
20. Unable or unwilling to complete the study procedures;
21. Patients that cannot be hospitalized in a radionuclide therapy room;
22. Patients with urinary incontinence;
23. Patients that are unable to comply with thyroid protective pre-medication;
24. Patients in whom bladder catheterization cannot be performed, or in patients who are unwilling to be catheterized if necessary;
25. Patients with contraindications for undergoing MRI or computed tomography (CT), including for receiving contrast agents; or
26. Patient is the Investigator or sub-Investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof, who is directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Delara, Study Director — Precirix
Locations (12):
- United States (9):
  - City of Hope, Duarte, California
  - Stanford University Medical Center, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Advanced Molecular Imaging & Therapy, Glen Burnie, Maryland
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
- Canada (3):
  - Princess Margaret Hospital, Toronto, Ontario
  - Hospital Notre Dame du CHUM, Montreal, Quebec
  - McGill University Faculty of Medicine - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Derived] D'Huyvetter M, Vos J, Caveliers V, Vaneycken I, Heemskerk J, Duhoux FP, Fontaine C, Vanhoeij M, Windhorst AD, Aa FV, Hendrikse NH, Eersels JLE, Everaert H, Gykiere P, Devoogdt N, Raes G, Lahoutte T, Keyaerts M. Phase I Trial of 131I-GMIB-Anti-HER2-VHH1, a New Promising Candidate for HER2-Targeted Radionuclide Therapy in Breast Cancer Patients. J Nucl Med. 2021 Aug 1;62(8):1097-1105. doi: 10.2967/jnumed.120.255679. Epub 2020 Dec 4. PMID 33277400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began in September 2021 and ended in May 2023. The majority of patients were recruited from major hospitals.
Pre-assignment Details: Patient 203-001 (Cohort 3) passed screening but was withdrawn prior to being administered study drug due to an SAE.
Groups:
- Cohort 1 CAM-H2 (2 x 1.85 GBq): Cohort 1: Patients will receive at least 1 cycle of CAM-H2 (2 x 1.85 GBq). Patients with CB may receive up to 4 cycles of CAM-H2, as long as the cumulative kidney dose remains <23 Gy (based on the dosimetry results during Cycle 1). Cycles will be given as 2 IV administrations, 4 weeks apart.
- Cohort 2 CAM-H2 (2 x 3.7) GBq: Cohort 2: Patients will receive at least 1 cycle of CAM-H2 (2 x 3.7 GBq). Patients with CB may receive up to 4 cycles of CAM-H2, as long as the cumulative kidney dose remains <23 Gy (based on the dosimetry results during Cycle 1). Cycles will be given as 2 IV administrations, 4 weeks apart.
- Cohort 3 CAM-H2 (2 x 5.55) GBq: Cohort 3: Patients will receive at least 1 cycle of CAM-H2 (2 x 5.55 GBq). Patients with CB may receive up to 4 cycles of CAM-H2, as long as the cumulative kidney dose remains <23 Gy (based on the dosimetry results during Cycle 1). Cycles will be given as 2 IV administrations, 4 weeks apart.
Period: Overall Study
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
Started (# of patients that passed screening and administered study drug) | 3 | 3 | 7
Completed | 1 | 1 | 3
Not Completed | 2 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Progressive Disease | 0 | 1 | 3
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq | Total
Number analyzed (Participants) | 3 | 3 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants] — Males and females greater than or equal to 18 years of age at screening
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 2 | 6 | 11
    >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 6 | 10
  Male | 0 | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 3 | 7 | 13
Weight [Mean (Full Range); unit: kg] | 52.8 [41.4 to 62] | 71.2 [59 to 80.5] | 73.3 [50 to 95.9] | 68.1 [41.4 to 95.9]
Baseline ECOG PS [Number; unit: participants] — ECOG score ranges from 0-5, lower ECOG scores indicate a higher likelihood of tolerating treatment and higher ECOG scores suggest greater disability and may indicate a poorer prognosis
  Scale:
  0: Able to carry on all pre-disease activities
  1. Restricted in strenuous activity but ambulatory and able to carry out light work
  2. Capable of all self-care but unable to carry out any work activities
  3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  5. Dead
  participants
    ECOG - 0 | 2 | 3 | 3 | 8
    ECOG - 1 | 1 | 0 | 4 | 5
Cancer Type [Number; unit: participants]
  Breast | 3 | 1 | 5 | 9
  Gastric | 0 | 1 | 1 | 2
  GEJ | 0 | 1 | 1 | 2
Brain Metastases Status [Number; unit: participants]
  Yes | 1 | 0 | 1 | 2
  No | 2 | 3 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT) Rate Within the First Cycle
Description: Dose-limiting toxicity (DLT) rate of CAM-H2 assessed by toxicities occurring within the first cycle
Time Frame: Within the first cycle of CAM-H2, up to 12 weeks
Population: Any Dose-Limiting Toxicities (DLTs) that occur during the first cycle by patients
Measure: Number; unit: DLTs
Groups:
- Cohort 1 CAM-H2 (2 x 1.85 GBq); Cohort 2 CAM-H2 (2 x 3.7) GBq; Cohort 3 CAM-H2 (2 x 5.55) GBq: Any Dose-Limiting Toxicities (DLTs) that occur during the first cycle
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
Number analyzed (Participants) | 3 | 3 | 7
DLTs | 0 | 0 | 1

2. Primary Outcome: Safety and Tolerability - Number of Treatment-emergent Adverse Events (TEAEs)
Description: Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: 18 months
Measure: Number; unit: Adverse Events
Groups:
- Cohort 1 CAM-H2 (2 x 1.85 GBq); Cohort 2 CAM-H2 (2 x 3.7) GBq; Cohort 3 CAM-H2 (2 x 5.55) GBq: Number of treatment-emergent adverse events (TEAEs)
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
Number analyzed (Participants) | 3 | 3 | 7
Adverse Events
  Grade 1 - Mild | 27 | 24 | 43
  Grade 2 - Moderate | 7 | 6 | 22
  Grade 3 - Severe | 2 | 3 | 8
  Grade 4 - Life-Threatening | 0 | 0 | 0
  Grade 5 - Death | 0 | 0 | 0

3. Secondary Outcome: To Assess the Clinical Benefit (CB) of CAM-H2
Description: Evaluate proportion of patients with a Complete Response, Partial Response, and Stable Disease in the dose escalation phase
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
Number analyzed (Participants) | 3 | 3 | 7
Participants
  Stable Disease (SD) | 1 | 0 | 2
  Progressive Disease (PD) | 2 | 3 | 4
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0
  Not Evaluable | 0 | 0 | 0
  Not Applicable (NA) - Stable disease less than 8 weeks | 0 | 0 | 1

4. Secondary Outcome: Anti-drug Antibodies (ADAs) Development
Description: Percentage of patients on CAM-H2 who develop anti-drug antibodies (ADAs)
Time Frame: 18 months
Population: Number of patients on CAM-H2 who develop anti-drug antibodies (ADAs)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 CAM-H2 (2 x 1.85 GBq): Cohort 1: Patients who had a positive ADA screen at ET/EOT that was confirmed positive for anti-CAMH-H2 antibodies
- Cohort 2 CAM-H2 (2 x 3.7) GBq: Cohort 2: Patients who had a positive ADA screen at ET/EOT that was confirmed positive for anti-CAMH-H2 antibodies
- Cohort 3 CAM-H2 (2 x 5.55) GBq: Cohort 3: Patients who had a positive ADA screen at ET/EOT that was confirmed positive for anti-CAMH-H2 antibodies
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
Number analyzed (Participants) | 3 | 3 | 7
Participants | 1 | 0 | 1

5. Secondary Outcome: Dosimetry Efficacy - Total Absorbed Dose
Description: Thirteen patients in 3 different dose levels were evaluated. The total absorbed dose for the 3 source organs (kidneys, liver, red marrow)
Time Frame: 18 months
Measure: Mean (Full Range); unit: Gy
Groups:
- Cohort 1 CAM-H2 (2 x 1.85 GBq); Cohort 2 CAM-H2 (2 x 3.7) GBq: Three patients were evaluated. The total absorbed dose for the 3 source organs (kidneys, liver, red marrow)
- Cohort 3 CAM-H2 (2 x 5.55) GBq: Seven patients were evaluated. The total absorbed dose for the 3 source organs (kidneys, liver, red marrow)
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
Number analyzed (Participants) | 3 | 3 | 7
Gy
  Kidney | 2.94 [2.05 to 3.47] | 4.68 [3.49 to 6.36] | 6.78 [1.45 to 11.27]
  Liver | 0.84 [0.52 to 1.28] | 1.62 [1.39 to 2.07] | 3.65 [0.88 to 6.46]
  Red Marrow | 0.30 [0.2 to 0.51] | 0.53 [0.42 to 0.60] | 0.95 [0.27 to 1.44]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from time signing informed consent through study completion, an average of 18 months
Groups:
- Cohort 3 CAM-H2 (2 x 5.55) GBq: Cohort 2: Patients will receive at least 1 cycle of CAM-H2 (2 x 5.55 GBq). Patients with CB may receive up to 4 cycles of CAM-H2, as long as the cumulative kidney dose remains <23 Gy (based on the dosimetry results during Cycle 1). Cycles will be given as 2 IV administrations, 4 weeks apart.
Arm/Group | Cohort 1 CAM-H2 (2 x 1.85 GBq) | Cohort 2 CAM-H2 (2 x 3.7) GBq | Cohort 3 CAM-H2 (2 x 5.55) GBq
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/3 | 3/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 CAM-H2 (2 x 1.85 GBq) (N=3) | Cohort 2 CAM-H2 (2 x 3.7) GBq (N=3) | Cohort 3 CAM-H2 (2 x 5.55) GBq (N=7)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 CAM-H2 (2 x 1.85 GBq) (N=3) | Cohort 2 CAM-H2 (2 x 3.7) GBq (N=3) | Cohort 3 CAM-H2 (2 x 5.55) GBq (N=7)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localized Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 2 (4) | 2 (3)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Urea Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (3) | 2 (2)
Fear of Falling (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Decrease Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid Margin Crusting (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04467515/Prot_SAP_001.pdf